CLINICAL TRIAL: NCT06902766
Title: Towards Digital Management of Pediatric Asthma:a Pilot Study
Brief Title: Towards Digital Management of Paediatric Asthma
Acronym: FrenchCare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP211434; ID-RCB Number:2022-A02649-34 (Other: ID-RCB Number:2022-A02649-34)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Asthma
Keywords: Pediatric asthma; Digital revolution; Digital inhaler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital medicine (Experimental): Active telemonitoring using real-time data from digital inhalers
  Interventions: Device: Active telemonitoring using real-time data from digital inhalers.
- Standardized medicine (Active Comparator): The patients are monitored as usual according to the standard care protocol. Patients will receive 2 digital inhalers, but only to record their treatment use.
  Interventions: Other: Standard

INTERVENTIONS:
Device: Active telemonitoring using real-time data from digital inhalers. — Telemonitoring system relying on the use of 2 digital inhalers FindAir ONE for pMDI, one for the controller the other for the reliever treatment.
  Active telemonitoring using real-time data from digital inhalers.
  Investigators will be alerted by email if a child:
  1. fails to take his or her controller treatment for 4 continuous days and/or
  2. uses > 4 doses of reliever treatment over 24 hours
  3. uses < 12 doses of reliever treatment over 3 months (indication to decrease the controller treatment)
  In these cases, investigators will be asked to schedule a teleconsultation within 2 working days with the family and to adapt treatments as needed. They may ask the family to use the portable spirometer and oximeter if necessary.
  No systematic consultation will be planned.
  Arms: Digital medicine
Other: Standard — Standardized care + passive recording of asthma treatment use (controller and reliever treatments) using digital inhalers
  Arms: Standardized medicine

SUMMARY:
This pilot study aims to explore whether a digital approach to managing childhood asthma using connected inhalers and video consultations triggered by alerts from these devices - could work as well as standard in-person care. The connected inhalers track when children use their daily prevention medication and their rescue medication for asthma symptoms. If a child misses several days of prevention medication or uses their rescue inhaler frequently, their doctor receives an alert and can schedule a video consultation to adjust their treatment. Fifty children aged 4-12 years with asthma will participate for 8 months, with half using this digital system and half receiving usual care. The study will measure whether this new approach is practical and acceptable to families and doctors, and will look at its effects on asthma control, quality of life, and healthcare use. The results will help design a larger study to fully test if this digital approach could improve asthma care for children.

DETAILED DESCRIPTION:
Asthma is the most common chronic illness in children. In France, two-thirds of children have uncontrolled asthma, meaning they experience symptoms and occasional asthma attacks.

The digital revolution has enabled the development of connected devices, particularly smart inhalers, which collect objective information for assessing asthma from patients' homes. The Covid-19 pandemic has further accelerated the adoption of telemedicine. These new approaches represent a significant shift in paediatric asthma management, offering opportunities for more effective treatment methods.

As a precursor to a larger investigation, this pilot study hypothesises that digital asthma management using proactive remote care through telemedicine consultations triggered by connected device alerts may improve childhood asthma control compared to current management approaches.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 to 12, whose asthma has been diagnosed by a physician
* Followed up for their asthma by a pediatrician or pediatric pulmonologist
* With asthma severity corresponding to GINA grades 2, 3 or 4 (Global Asthma Initiative Guidelines)
* Whose controller and reliever treatments are administered using pressurized metered-dose inhalers (p-MDIs)
* With social security
* Whose parents or legal guardian(s):

  * Have given their written and informed consent for their child's participation and their participation,
  * Have a smartphone in the household that can download the application and is compatible with it,
  * Are capable, in the opinion of the investigator, of understanding the use of the mobile application and module FRENCH CARE specifically dedicated to the research and the digital inhalers provided.

Non-inclusion Criteria:

* Patients with another pathology that could interfere with the evaluation of the endpoints (e.g, bronchopulmonary dysplasia, cystic fibrosis, etc.)
* Patients whose parents or legal representative(s) are, in the opinion of the investigator, unable to understand the purpose of the study and/or express their consent.
* Patients benefiting from State Medical Aid

Exclusion Criteria:

- Patient who did not use the system within 15 days of the inclusion visit

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in asthma severity measured by the Composite Asthma Severity Index (CASI) | At the inclusion visit (baseline) and 8 months (+/- 1 month) (end of study) in each group
  The CASI is a validated composite score that evaluates asthma severity by incorporating measures of asthma symptoms, exacerbations, lung function, and treatment level. The change in CASI score will be compared between groups, calculated as the difference between the final score (at 8 months) and the baseline score. Lower scores indicate less severe asthma.
  The CASI ranges from 0 to 17, with higher scores meaning a higher severity (worse outcome).

SECONDARY OUTCOMES:
Asthma control | At the inclusion visit (baseline) and 8 months (+/- 1 month) (end of study) in each group
  Evolution in the overall Childhood Asthma Control Test (c-ACT) score. The c-ACT (Childhood Asthma Control Test) will be used to evaluate the evolution of asthma control.
  The c-ACT ranges from 0 min to 27 max, with higher scores meaning better asthma control (better outcome).
Severe exacerbations requiring oral steroids | During the eight-month follow up period in each group
  Severe exacerbations (defined as an exacerbation requiring oral corticosteroid therapy): number of severe exacerbations per patient and percentage of patients with at least one severe exacerbation
Severe exacerbations requiring emergency department visit and/or hospital admission. | During the eight-month follow up period in each group
  Severe exacerbations requiring emergency department visits and/or hospitali admission: number per patient and percentage of patients with at least one
Children's lung function | At the inclusion visit (baseline) and 8 months (+/- 1 month) (end study) in each group
  Evolution of lung function assessed by the predicted percentage of the forced expiratory volume in one second (FEV1) in children aged 7 to 12 years
Quality of life questionnaire | At the inclusion visit (baseline) and 8 months (+/- 1 month) (end of study) in each group
  Children (aged 7 -12 years) were assessed by the mini Pediatric Asthma Quality of Life Questionnaire (mPAQLQ). Their parents were assessed by the Pediatric Asthma Caregivers' Quality of Life.
Adherence | During the eight-month follow up period in each group
  The adherence of patients to their maintenance treatment, automatically recorded via digital inhalers, defined as the number of doses taken divided by the number of doses prescribed x 100: average percentage of adherence
Reliever treatment | During the eight-month follow up period in each group
  Use of reliever treatment (salbutamol) is automatically recorded via digital inhalers: average number of uses per each patient
Number of teleconsultations/consultations | During the eight-month follow up period in each group
  Average number of consultations/teleconsultations per patient, scheduled and unscheduled, and their average cumulative duration per patient
Children participation | During the eight-month follow up period in each group
  The child's speaking time compared to the total speaking time (child + parent + doctor), expressed as a percentage was determined from video recordings.
  The number of the child's speech turns compared to the total number of speech turns (child + parent + doctor), expressed as a percentage.
  The number of complete thoughts, or "utterances", of the child compared to the total number of complete thoughts, expressed as a percentage.
  The child's non-verbal communication, analyzed by a module of the Roter Interactive Assessment System
Absenteeism | During the eight-month follow up period in each group
  Number of days of asthma-related absenteeism (from school for children and work for parents), per patient
Satisfaction of parents | After 8 months (+/- 1 month) (end of study)
  Assessed by the proportion of parents in the experimental group responding on a custom questionnaire that they wish to continue the digital management experience and the reason for their choice
Satisfaction of doctors | After 8 months (+/- 1 month) (end of study)
  Assessed by the proportion of doctors in the experimental group responding on a custom questionnaire that they wish to continue the digital management experience and the reason for their choice

CONTACTS AND LOCATIONS:
Overall Officials: David DUMMOND, MD, PhD, Principal Investigator — Hôpital Necker Enfants Malades AP-HP
Locations (1):
- Hôpital Necker Enfants Malades AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No